CLINICAL TRIAL: NCT01874652
Title: Assessment of Safety & Efficacy of Light Weight Breast Implant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0007-13-BNZ
Record Dates: First submitted 2013-05-23; First posted 2013-06-11 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2014-12

CONDITIONS: Breast Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Light Weight Breast Implants (Experimental): Assessment of Safety and Efficacy of Light Weight Breast Implant
  Interventions: Device: Light Weight Breast Implants

INTERVENTIONS:
Device: Light Weight Breast Implants — Light Weight Breast Implants

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of Light Weight Breast Implant (LWBI) in breast augmentation.

DETAILED DESCRIPTION:
This is a Single-center. The purpose of the study is to evaluate safety and effectiveness of LWBI in breast augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Genetic women at ages 18 to 65 seeking breast enlargement
* Signed informed consent
* Agreement to complete all required follow up visits
* A medically acceptable candidate
* Sufficient breast tissue for proper implant coverage (≥20 mm by pinch test)

Exclusion Criteria:

* Patients with active infection anywhere in their body
* Women who are currently pregnant or nursing
* Insufficient tissue covering in the prospective area of implantation (e.g. after preceding breast reduction), radiation damage or reduced vascularization
* Abscesses, malignant tumors(cancer or recurrent metastases), advanced fibrocystic diseases
* Patients with a history of psychiatric treatment
* Patients that been implanted with any silicone implant (e.g. silicone artificial joints, facial implants)
* Expected allergies or extraordinary immune response to implants
* Wound healing impairments or heavy burn scars
* Existing costal injuries
* The Patient Participated in an investigational trial within 30 days of enrollment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
No reoperation | during 6 months follow up period

SECONDARY OUTCOMES:
Duration for all adverse events (AEs) on per patient and per implant basis will be recorded and analyzed. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Noam Calderon, md, Principal Investigator — Bnai-Zion
Locations (1):
- Bnai Zion, Haifa, Israel